CLINICAL TRIAL: NCT06687005
Title: Comparative Analysis of Gremlin-1, Syndecan-4 and IL-1 Beta Levels in Gingival Crevicular Fluid Among İndividuals With Periodontal Health and Stage III Periodontitis, Considering Both Smokers and Non-Smokers, Before and After Non-Surgical Periodontal Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Tugba Aydin (Other)
Responsible Party: Sponsor-Investigator, Tugba Aydin, TAYdin, Ataturk University
Organization: Ataturk University (Other)
Other Study IDs: 2024/01-16
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Periodontitis (Stage 3); Gremlin-1; Syndecan 4; Interleukin 1-beta
MeSH Terms: conditions — Periodontitis; Polyposis Syndrome, Hereditary Mixed, 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers with stage 3 periodontitis
  Interventions: Procedure: non-surgical periodontal therapy
- Non-smokers with stage 3 periodontitis
  Interventions: Procedure: non-surgical periodontal therapy
- Healthy Participant

INTERVENTIONS:
Procedure: non-surgical periodontal therapy — non-surgical periodontal therapy
  Groups: Non-smokers with stage 3 periodontitis; Smokers with stage 3 periodontitis

SUMMARY:
eriodontitis is a complex disease characterized by the inflammation and destruction of the tissues supporting the teeth, and smoking can adversely affect the pathophysiological changes in this process. In an unhealthy periodontium, the host's inflammatory response products can be detected in the content of DOS, and the presence of these components is crucial in obtaining information about the pathogenesis of periodontal disease. Biochemical markers found in DOS are significantly helpful in determining the active stages and regions of the disease and in evaluating the host response to periodontal treatment. IL-1β has been determined to play a leading role in the pathogenic mechanism of periodontal tissue destruction, and the degree of inflammation in the tissues can be measured by IL-1β activity in DOS. Syndecan-4, a member of the transmembrane heparan sulfate proteoglycan family, regulates cellular activities such as tissue homeostasis, inflammation, fibrosis, and tumor metastasis. Gremlin-1 is a protein that inhibits BMP (Bone Morphogenetic Protein) signaling, influencing cell growth and tissue development. Gremlin-1 plays an important role in tissue repair and regeneration, modulating inflammatory processes and regulating cellular homeostasis. While recent studies have explained the role of Syndecan-4 and Gremlin-1 in inflammation, their effects on periodontal tissues are still quite limited in the literature. Our study aims to investigate the effects of smoking on these biomarkers by comparing the periodontal status before and after treatment of healthy, smoking, and non-smoking individuals with stage 3 periodontitis, with the goal of developing early diagnostic tools in the future.

DETAILED DESCRIPTION:
Periodontal diseases are inflammatory conditions that affect a significant portion of the global population. The cleaning of supragingival and subgingival dental calculus and flap surgery when necessary are treatment options. If left untreated, they lead to the loss of teeth and the supporting tissues. Numerous bacterial species colonize the oral cavity and can alter the delicate balance between the host and bacteria in the development of periodontal disease. While it begins with subgingival microbial plaque, the origin of periodontitis is based on the tissue destruction mediators produced by the host response to pathogenic infections. Periodontitis is classified into stages and grades according to the severity and progression of the disease. In stage III periodontitis, significant interdental clinical attachment loss (CAL) is observed, and in the absence of treatment, tooth loss may occur. This stage is characterized by bone destruction extending to the middle of the tooth root, bone intrabony pockets, and periodontal lesions. Class II or III furcation involvement may also be observed. To diagnose a patient with stage III periodontitis, the interdental CAL must be greater than 5 mm, the tooth loss due to periodontitis should be fewer than four teeth, and the probing pocket depth (PPD) should be ≥6 mm, with at least 3 mm vertical bone loss. The goal of periodontal treatment is to maintain and restore the health of the tissues surrounding and supporting the teeth. Due to the accumulation of cement, plaque, and calculus within the periodontal pocket, the surface becomes contaminated by bacteria and enzymes. Nonsurgical periodontal therapy is a frequently used method for the treatment of periodontitis. The main aim is to remove microbial biofilm from the diseased root surface without surgical intervention and without removing the surrounding soft tissue. In this way, the diseased root surface is biologically compatible, supporting the reattachment of periodontal tissues to the tooth. The analysis of Gingival Crevicular Fluid (GCF) is a sensitive diagnostic approach in studying the host's activity in periodontal diseases. In an unhealthy periodontium, the host's inflammatory response products can be detected in the content of GCF, and the presence of these components is crucial for obtaining information about the pathogenesis of periodontal disease. Biochemical evaluation of GCF is important not only for the early detection of periodontal disease but also for showing associations with connective tissue destruction products and bone metabolism. The biochemical markers in GCF are significantly helpful in determining the active stages and regions of the disease and in evaluating the host response to periodontal treatment. IL-1β plays a pioneering role in the pathogenic mechanism of periodontal tissue destruction. The severity of periodontal disease can be determined by the activity of this cytokine. According to studies, clinical parameters such as Gingival Index (GI) and Probing Pocket Depth (PPD) are correlated with IL-1β activity in GCF. The intensity of inflammation in periodontal tissues can be measured by IL-1β activity in GCF. Smoking has been shown in studies to have negative effects on oral health, as it does on general health. In individuals who smoke, periodontal diseases tend to be more common and severe. Smoking has been shown to increase inflammation in periodontal tissues, negatively affect tissue healing, and suppress the immune system. In this context, the effects of smoking on the treatment outcomes of patients with periodontitis should be studied in detail. Syndecan-4, a member of the transmembrane heparan sulfate proteoglycan family, binds to extracellular effector molecules and regulates cellular processes such as tissue homeostasis, inflammation, fibrosis, and tumor metastasis. Due to its ability to regulate cell adhesion, modulate signal transduction, and influence cell migration, Syndecan-4 plays a critical role in cell behavior and tissue organization. Gremlin-1, one of the antagonists of bone morphogenetic proteins (BMPs), contains a cysteine knot and is a member of the cysteine knot superfamily. Gremlin-1 is a protein that inhibits BMP signaling and is a factor influencing cell growth and tissue development. Gremlin-1 plays an important role in tissue repair and regeneration, modulating inflammation processes and regulating cellular homeostasis. The changes in Syndecan-4 levels and their impact on periodontal health under smoking and periodontitis conditions should be studied to better understand the role of this molecule in periodontal disease. Understanding how Gremlin-1 levels change in patients with periodontitis and smokers can contribute to a better understanding of periodontal health and the development of more effective treatment strategies. In the planned study, the changes in the levels of Gremlin-1, Syndecan-4, and IL-1β in periodontitis, a significant disease of oral and dental health, will be investigated to provide new information to the literature.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers must not have any systemic diseases.
* The volunteers must be between 18 and 60 years of age.
* Control group: Periodontally healthy patients with no signs of periodontal disease and no history of smoking.
* Study Group I: Non-smoking patients with stage III periodontitis, evaluated based on clinical findings such as PD ≥ 5 mm and CAL ≥ 4 mm (with ≥ 30% of affected teeth), without radiographic evidence of bone loss and a history of smoking.
* Study Group II: Smoking patients with untreated stage III periodontitis, evaluated based on clinical findings such as PD ≥ 5 mm and CAL ≥ 4 mm (with ≥ 30% of affected teeth), with radiographic evidence of bone loss and a history of smoking for at least 10 cigarettes per day over the past 3 years.

Exclusion Criteria:

* The individual's unwillingness to participate in the study
* Being outside the specified age range
* Pregnant or breastfeeding patients
* Having a systemic disease
* Smoking in the past 10 years
* Having received periodontal treatment within the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include a total of 45 volunteer individuals, consisting of 15 smokers and 15 non-smokers diagnosed with stage 3 periodontitis, aged 18-60, who seek treatment for periodontal complaints such as pain, sensitivity, and gum recession at the Department of Periodontology, Faculty of Dentistry, Atatürk University, as well as 15 healthy individuals. The sampling procedure will be carried out at the Department of Periodontology, Faculty of Dentistry, Atatürk University, with the approval of the ethical committee report from the Scientific Research Ethics Committee of Erzurum Medical Faculty.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
assesment of Gremlin-1 pre-treatment | From enrollment to the end of treatment at 3 months
  Measurement of Gremlin-1 levels using an ELISA kit from gingival crevicular fluid samples taken from patients before periodontitis treatment.
assesment of syndecan-4 pre treatment | From enrollment to the end of treatment at 3 months
  Measurement of Syndecan-4- levels using an ELISA kit from gingival crevicular fluid samples taken from patients before periodontitis treatment.
Assesment of IL-1 Beta pre-treatment | From enrollment to the end of treatment at 3 months
  Measurement of IL-1 Beta levels using an ELISA kit from gingival crevicular fluid samples taken from patients before periodontitis treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes